CLINICAL TRIAL: NCT05362110
Title: A Multicenter, Randomized, Double-blind, Phase 3 Study to Evaluate Efficacy and Safety of HCP1803 in Patients With Essential Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of HCP1803 in Patients With Essential Hypertension
Acronym: HM_APOLLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-APOLLO-301
Record Dates: First submitted 2022-05-01; First posted 2022-05-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): HCP1803-3
  Interventions: Drug: HCP1803-3; Drug: HPP2004
- Active Comparator (Active Comparator): RLD2002
  Interventions: Drug: RLD2002; Drug: HPP2003-3

INTERVENTIONS:
Drug: HCP1803-3 — Take it once daily for 8 weeks orally.
  Arms: Experimental
Drug: RLD2002 — Take it once daily for 8 weeks orally.
  Arms: Active Comparator
Drug: HPP2003-3 — Placebo drug. Take it once daily for 8 weeks orally.
  Arms: Active Comparator
Drug: HPP2004 — Placebo drug. Take it once daily for 8 weeks orally.
  Arms: Experimental

SUMMARY:
A multicenter, randomized, double-blind, phase 3 study to evaluate efficacy and safety of HCP1803 in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension whose blood pressure measured in visit1 corresponds to the following conditions

   * mean sitSBP <180 mmHg and mean sitDBP < 110 mmHg for patients receiving any BP-lowering drug within 1 month prior to Visit 1
   * 140 mmHg ≤ mean sitSBP < 180 mmHg and 60 mmHg ≤ mean sitDBP < 110 mmHg for patients not receiving BP-lowering drugs within 1 month prior to Visit 1
2. Patients with essential hypertension who meet 140 mmHg ≤ mean sitSBP < 180 mmHg and 60 mmHg ≤ mean sitDBP < 110 mmHg at Visit 2

Exclusion Criteria:

1. Difference between arms greater than 20 mmHg for mean sitSBP or 10 mmHg for mean sitDBP at Visit 1
2. Orthostatic hypotension with symptoms within 3 months prior to visit 1.
3. Secondary hypertensive patient or suspected to be
4. Uncontrolled diabetes mellitus(HbA1c > 9%) or type I diabetes mellitus
5. Active gout or hyperuricemia (uric acid ≥ 9mg/dL)
6. Severe heart disease or severe neurovascular disease
7. Moderate or malignant retinopathy
8. Clinically significant hematological finding
9. Severe renal diseases (eGFR<30mL/min/1.73m2)
10. Severe or active hepatopathy (AST or ALT ≥ 3 times of normal range)
11. Hypokalemia or Hyperkalemia(K<3.5mmol/L or K ≥ 5.5mmol/L)
12. Hyponatremia or Hypernatremia(Na<135mmol/L or Na ≥ 155mmol/L)
13. Hypercalcemia
14. History of malignancy tumor
15. History of autoimmune disease
16. History of alcohol or drug abuse
17. Positive to pregnancy test, nursing mother, intention on pregnancy
18. Considered by investigator as not appropriate to participate in the clinical study with other reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic blood pressure | baseline, 8 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting systolic blood pressure | baseline, 4 weeks
Change from baseline in sitting distolic blood pressure | baseline, 4 weeks, 8 weeks
Proportion of subjects achieving blood pressure control | 4 weeks, 8 weeks
Blood pressure response rate | 4 weeks, 8 weeks
Treatment response rate | 4 weeks, 8 weeks
Change from baseline in pulse pressure | baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, M.D., Ph.D., Principal Investigator — Donggguk University Ilsan Hospital
Locations (1):
- Donggguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No